CLINICAL TRIAL: NCT04033107
Title: Clinical Research of High Dose Vitamin C Combined With Metformin in the Treatment of Malignant Tumors
Brief Title: High Dose Vitamin C Combined With Metformin in the Treatment of Malignant Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Zhou Fuxiang, Principal Investigator, Clinical Professor, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZNCM
Record Dates: First submitted 2019-07-20; First posted 2019-07-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hepatocellular Cancer; Pancreatic Cancer; Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Colorectal Neoplasms | interventions — Ascorbic Acid; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Vitamin C combined with metformin
  Interventions: Drug: Vitamin C; Drug: Metformin

INTERVENTIONS:
Drug: Vitamin C — Participants will receive intravenous Vitamin C injection (dose: 1.5g/kg, D1-3, every 2 weeks), treatment termination when the disease progress is confirmed.
  Other Names: Ascorbic acid
Drug: Metformin — Participants will orally take metformin 4g daily.

SUMMARY:
This is an open, prospective, single-arm, multi-cohort clinical study to evaluate the efficacy and safety of high-dose vitamin C combined with metformin in the treatment of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years to 75 years.
2. Had a disease status that was measurable or evaluable as defined by Response Evaluation Criteria in Solid Tumors (RECIST, version1.1)： Cohort A: patients with advanced hepatocellular carcinoma who had failed previous standard first-line therapy and could not tolerate or reject existing therapies.

   Cohort B: patients with advanced pancreatic cancer who had previously failed standard first-line therapy, could not tolerate or reject existing therapies.

   Cohort C: patients with advanced gastric cancer who had failed previous standard second-line or above treatment, who could not tolerate or reject existing therapies.

   Cohort D: patients with advanced colorectal cancer who had failed previous standard second-line or above treatment, who could not tolerate or reject existing therapies.
3. Adequate hepatic, renal, heart, and hematologic functions (hemoglobin ≥80g/L, platelets ≥ 80×10^9/L, neutrophils ≥ 1.5×10^9/L, total bilirubin within 1.5×the upper limit of normal(ULN), ALT and AST≤2.5×the ULN (If liver metastases, serum transaminase≤5×the ULN), serum creatine ≤ 1.5 x ULN, creatinine clearance rate > 50ml/min).
4. At least 4 weeks after the last anti-tumor treatment (surgery, chemotherapy, radiotherapy, biotherapy or endocrine therapy) before enrollment.
5. Had a life expectancy of at least 3 months.
6. Had an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2.
7. Signed informed consent.

Exclusion Criteria:

1. In the past or at the same time with other malignant tumors (already cure period of IB or cervical, lower levels of noninvasive basal cell or squamous cell cancer, obtain complete remission (CR) > 10 years of breast cancer, obtain complete remission (CR) > 10 years of malignant melanoma, obtain complete remission (CR) > 5 years except of other malignant tumors).
2. Pregnant or lactating female patients.
3. Those who have applied excessive dose of vitamin C or (and) metformin in recent 1 month.
4. Patients with glucose-6-phosphate dehydrogenase deficiency.
5. Patients with hydronephrosis.
6. Had a history of clinically significant or uncontrolled heart disease, including but not limited to: (1)Myocardial infarction. (2)Angina.(3)Congestive heart failure above grade 2 of the New York heart association (NYHA).(4)Ventricular arrhythmias requiring continuous treatment.(5)Supraventricular arrhythmias, including uncontrolled atrial fibrillation.
7. The patients had mental disorders, and the researchers believed that the patients could not fully or fully understand the possible complications in this study.
8. Have a history of immunodeficiency, including: HIV positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation.
9. Those who cannot tolerate or may be allergic to the drugs used in this study.
10. Participated in clinical trials of other drugs within the past 1 month.
11. Other factors considered unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 12 weeks
  Defined as time from first dose of treatment to death from any cause, or even radiological detection/or clinical of disease progression.

SECONDARY OUTCOMES:
Overall survival | up to 12 weeks
  Defined as time from first dose of treatment until death.
Objective response rate | up to 12 weeks
  Overall Response Rate, as determined by the percentage of patients achieving Partial or Complete response per RECIST 1.1.
Disease control rate | up to 12 weeks
  Disease Control Rate: the number of patients with a CR, PR or SD lasting at least 2 months per RECIST 1.1.
Changes of quality of life | up to 12 weeks
  Examination of quality of life by EORTC QLQ-C30 questionnaire every 8 weeks.
Number of participants with treatment-related adverse events as assessed by CTCAE v3.0 | up to 12 weeks
  The number of grade 1-4 and grade 5 (fatal) NCI Common Terminology Criteria for Adverse Events Version 3.0 (CTCAE) events during treatment. All patients will be evaluable for toxicity from the time of their first treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fuxiang Zhou, M.D, Study Chair — Wuhan University
Locations (1):
- Zhongnan Hopital of Wuhan University, Wuhan, Hubei, China